CLINICAL TRIAL: NCT04608825
Title: Intensive Care Unit Management After Cardiac ARrest in Russia. - a Retrospective Observational Multi-center Cohort Study
Brief Title: Intensive Care Unit Management After Cardiac ARrest in Russia
Acronym: ICAR-RUS
Status: Completed | Type: Observational
Sponsor: Russian Federation of Anesthesiologists and Reanimatologists (Other)
Responsible Party: Sponsor
Other Study IDs: FARCT0003
Record Dates: First submitted 2020-10-21; First posted 2020-10-29 (Actual); Last update posted 2025-02-04 (Actual); Status verified 2025-01

CONDITIONS: Post Cardiac Arrest Syndrome
MeSH Terms: conditions — Post-Cardiac Arrest Syndrome

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
The purpose of this study is to study the prevalence of post cardiac arrest syndrome (PCAS) among ICU patients, to analyze the effectiveness of intensive care, to assess the factors associated with death and the development of severe neurological deficits.

DETAILED DESCRIPTION:
According to statistics, more than half of patients who have undergone cardiopulmonary resuscitation (CPR) die from acute cardiovascular or cerebral insufficiency caused by global ischemia. The survival rate after cardiac arrest and successful CPR is about 10%, with good neurological recovery from 0.9% to 7.8%.

The most common cause of cardiac arrest is heart failure, followed by respiratory failure. Despite progress in the provision of specialized medical care, the proportion of patients who underwent post cardiac arrest syndrome (PCAS) and discharged from the hospital remains very low, and neurological and mental disorders persist forever.

The prevalence of nosocomial cardiac arrest in adults varies, with an average of 6 to 9 cases per 1000 hospitalizations. The prevalence of nosocomial cardiac arrest in adults varies, with an average of 6 to 9 cases per 1000 hospitalizations. About half of inpatient cardiac arrests occur in specialized wards, and the remaining half in other locations, such as intensive care units (ICU) and operating rooms. Common causes of cardiac arrest include coronary artery disease, pulmonary embolism, poisoning with cardiotoxic agents (drugs, antidepressants, cardiac glycosides), metabolic disorders (most often hypo- or hyperkalemia), and sepsis.

Modern methods of intensive care of PCAS provide good results, but require significant diagnostic, therapeutic, human and economic resources. The recommendations of the European Resuscitation Council and the European Intensive Care Society on post-resuscitation care have had an impact on improving the quality of care. In Russia, such recommendations are not accepted. One of the conditions for the development and implementation of methods aimed at increasing the survival rate of patients with PCAS is the collection of up-to-date information on the prevalence, causes and patterns of the development of the disease.

In recent years In Russia, not a single multicenter study has been published on the statistics of survival after cardiac arrest and the results of intensive care. There is also no single algorithm for the treatment of post cardiac arrest syndrome, with the exception of the organ donation protocol; meanwhile, the majority of patients suffering from severe multiple organ failure in the postresuscitation period cannot be donors and die as a result of the progression of multiple organ failure.

Targeted therapy for PCAS includes respiratory and hemodynamic support, temperature management, laboratory monitoring, and anticonvulsant therapy. Predicting the degree of neurocognitive dysfunction remains a clinically difficult issue.

The study of PCAS is undoubtedly relevant and can help identify a number of additional prognostic factors affecting the outcome of the disease.

The purpose of this study is to examine the prevalence of PCAS in Russia, to analyze the effectiveness of intensive care methods, to evaluate the factors associated with death and the development of severe neurological deficits. Research centers are located on the intensive care units. A multicenter retrospective registry cohort study is planned.

The research centers are located on the basis of the ICU, of the Irkutsk Regional Clinical Hospital, Irkutsk City Clinical Hospital No.1, City Clinical Hospital No.3, Irkutsk; Federal research and clinical center of intensive care medicine and rehabilitology, Moscow; Orenburg regional clinical hospital, Orenburg City N.I. Pirogov Clinical Hospital, Orenburg; Kuzbass Clinical Emergency Hospital named after M.A. Podgorbunsky, Kemerovo; Regional clinical hospital, Krasnoyarsk interdistrict clinical hospital of emergency medical care named after NS Karpovich, Krasnoyarsk interdistrict clinical hospital №20 named after I.S. Berzona, Krasnoyarsk interdistrict clinical hospital №4, Krasnoyarsk.

Against the background of the assessment of vital functions, methods of respiratory support, laboratory data, and drug therapy will be compared. Continuous data will be presented as the median and interquartile range for the nonparametric distribution and as the mean and standard deviation for the parametric distribution. The categorical variables will be presented as the number of patients and the percentage of the total number of patients. For record keeping, an individual registration card.

ELIGIBILITY:
Inclusion Criteria:

* patients with out-of-hospital and in-hospital successful CPR; ·
* age - from 18 years old; ·
* survival after CPR - more than 24 hours.

Exclusion Criteria:

* age less than 18 years; ·
* death occurring less than 24 hours after CPR; ·
* oncological pathology in the terminal stage; ·
* severe neurological deficits and cognitive dysfunction that occurred before CPR.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients in ICU
Sampling Method: Non-Probability Sample
Enrollment: 500 (Actual)
Dates: Start 2020-05-11 (Actual); Primary Completion 2023-11-11 (Actual); Study Completion 2023-12-11 (Actual)

PRIMARY OUTCOMES:
incidence of PCAS in the ICU | during each patient hospitalization, an average of 1 month
  post cardiac arrest syndrome in patients of intensive care unit

CONTACTS AND LOCATIONS:
Overall Officials: Vladimir Gorbachev, MD, Principal Investigator — CEO Irkutsk State Medical Academy of Postgraduate Education
Locations (11):
- Russia (11):
  - CEO Irkutsk State Medical Academy of Postgraduate Education - Branch Campus of the FSBEI FPE RMACPE MOH Russia, Irkutsk
  - City Clinical Hospital No.3, Irkutsk
  - Irkutsk City Clinical Hospital No.1, Irkutsk
  - Kuzbass Clinical Emergency Hospital named after M.A. Podgorbunsky, Kemerovo
  - Krasnoyarsk interdistrict clinical hospital of emergency medical care named after NS Karpovich, Krasnoyarsk
  - Krasnoyarsk interdistrict clinical hospital №20 named after I.S. Berzona Krasnoyarsk, Russia, Krasnoyarsk
  - Krasnoyarsk interdistrict clinical hospital №4 Krasnoyarsk, Russia, Krasnoyarsk
  - Regional clinical hospital, Krasnoyarsk
  - Federal research and clinical center of intensive care medicine and rehabilitology, Moscow
  - Orenburg City N.I. Pirogov Clinical Hospital, Orenburg
  - Orenburg regional clinical hospital, Orenburg

REFERENCES:
- [Background] Andersen LW, Holmberg MJ, Berg KM, Donnino MW, Granfeldt A. In-Hospital Cardiac Arrest: A Review. JAMA. 2019 Mar 26;321(12):1200-1210. doi: 10.1001/jama.2019.1696. PMID 30912843
- [Background] Benjamin EJ, Blaha MJ, Chiuve SE, Cushman M, Das SR, Deo R, de Ferranti SD, Floyd J, Fornage M, Gillespie C, Isasi CR, Jimenez MC, Jordan LC, Judd SE, Lackland D, Lichtman JH, Lisabeth L, Liu S, Longenecker CT, Mackey RH, Matsushita K, Mozaffarian D, Mussolino ME, Nasir K, Neumar RW, Palaniappan L, Pandey DK, Thiagarajan RR, Reeves MJ, Ritchey M, Rodriguez CJ, Roth GA, Rosamond WD, Sasson C, Towfighi A, Tsao CW, Turner MB, Virani SS, Voeks JH, Willey JZ, Wilkins JT, Wu JH, Alger HM, Wong SS, Muntner P; American Heart Association Statistics Committee and Stroke Statistics Subcommittee. Heart Disease and Stroke Statistics-2017 Update: A Report From the American Heart Association. Circulation. 2017 Mar 7;135(10):e146-e603. doi: 10.1161/CIR.0000000000000485. Epub 2017 Jan 25. No abstract available. Erratum In: Circulation. 2017 Mar 7;135(10):e646. doi: 10.1161/CIR.0000000000000491. Circulation. 2017 Sep 5;136(10):e196. doi: 10.1161/CIR.0000000000000530. PMID 28122885
- [Background] Chan PS, McNally B, Tang F, Kellermann A; CARES Surveillance Group. Recent trends in survival from out-of-hospital cardiac arrest in the United States. Circulation. 2014 Nov 18;130(21):1876-82. doi: 10.1161/CIRCULATIONAHA.114.009711. PMID 25399396
- [Background] Chan PS, Nallamothu BK, Krumholz HM, Spertus JA, Li Y, Hammill BG, Curtis LH; American Heart Association Get with the Guidelines-Resuscitation Investigators. Long-term outcomes in elderly survivors of in-hospital cardiac arrest. N Engl J Med. 2013 Mar 14;368(11):1019-26. doi: 10.1056/NEJMoa1200657. PMID 23484828
- [Background] Dellinger RP, Levy MM, Rhodes A, Annane D, Gerlach H, Opal SM, Sevransky JE, Sprung CL, Douglas IS, Jaeschke R, Osborn TM, Nunnally ME, Townsend SR, Reinhart K, Kleinpell RM, Angus DC, Deutschman CS, Machado FR, Rubenfeld GD, Webb S, Beale RJ, Vincent JL, Moreno R; Surviving Sepsis Campaign Guidelines Committee including The Pediatric Subgroup. Surviving Sepsis Campaign: international guidelines for management of severe sepsis and septic shock, 2012. Intensive Care Med. 2013 Feb;39(2):165-228. doi: 10.1007/s00134-012-2769-8. Epub 2013 Jan 30. PMID 23361625
- [Background] Deye N, Cariou A, Girardie P, Pichon N, Megarbane B, Midez P, Tonnelier JM, Boulain T, Outin H, Delahaye A, Cravoisy A, Mercat A, Blanc P, Santre C, Quintard H, Brivet F, Charpentier J, Garrigue D, Francois B, Quenot JP, Vincent F, Gueugniaud PY, Mira JP, Carli P, Vicaut E, Baud FJ; Clinical and Economical Impact of Endovascular Cooling in the Management of Cardiac Arrest (ICEREA) Study Group. Endovascular Versus External Targeted Temperature Management for Patients With Out-of-Hospital Cardiac Arrest: A Randomized, Controlled Study. Circulation. 2015 Jul 21;132(3):182-93. doi: 10.1161/CIRCULATIONAHA.114.012805. Epub 2015 Jun 19. PMID 26092673
- [Background] Dragancea I, Rundgren M, Englund E, Friberg H, Cronberg T. The influence of induced hypothermia and delayed prognostication on the mode of death after cardiac arrest. Resuscitation. 2013 Mar;84(3):337-42. doi: 10.1016/j.resuscitation.2012.09.015. Epub 2012 Sep 20. PMID 23000363
- [Background] Elmer J, Scutella M, Pullalarevu R, Wang B, Vaghasia N, Trzeciak S, Rosario-Rivera BL, Guyette FX, Rittenberger JC, Dezfulian C; Pittsburgh Post-Cardiac Arrest Service (PCAS). The association between hyperoxia and patient outcomes after cardiac arrest: analysis of a high-resolution database. Intensive Care Med. 2015 Jan;41(1):49-57. doi: 10.1007/s00134-014-3555-6. Epub 2014 Dec 4. PMID 25472570
- [Background] Grasner JT, Meybohm P, Lefering R, Wnent J, Bahr J, Messelken M, Jantzen T, Franz R, Scholz J, Schleppers A, Bottiger BW, Bein B, Fischer M; German Resuscitation Registry Study Group. ROSC after cardiac arrest--the RACA score to predict outcome after out-of-hospital cardiac arrest. Eur Heart J. 2011 Jul;32(13):1649-56. doi: 10.1093/eurheartj/ehr107. Epub 2011 Apr 22. PMID 21515626
- [Background] Jakkula P, Reinikainen M, Hastbacka J, Loisa P, Tiainen M, Pettila V, Toppila J, Lahde M, Backlund M, Okkonen M, Bendel S, Birkelund T, Pulkkinen A, Heinonen J, Tikka T, Skrifvars MB; COMACARE study group. Targeting two different levels of both arterial carbon dioxide and arterial oxygen after cardiac arrest and resuscitation: a randomised pilot trial. Intensive Care Med. 2018 Dec;44(12):2112-2121. doi: 10.1007/s00134-018-5453-9. Epub 2018 Nov 14. PMID 30430209
- [Background] Zylke JW. Drug war intelligence gathering: risky, but useful to physicians. JAMA. 1988 Oct 21;260(15):2169-70. No abstract available. PMID 3172392
- [Background] Capani F, Della Loggia F, Sensi S. [Pancreatic diabetes. Diagnosis and therapy]. Minerva Med. 1976 Jan 28;67(4):301-6. No abstract available. Italian. PMID 1250522
- [Background] Lemiale V, Dumas F, Mongardon N, Giovanetti O, Charpentier J, Chiche JD, Carli P, Mira JP, Nolan J, Cariou A. Intensive care unit mortality after cardiac arrest: the relative contribution of shock and brain injury in a large cohort. Intensive Care Med. 2013 Nov;39(11):1972-80. doi: 10.1007/s00134-013-3043-4. Epub 2013 Aug 14. PMID 23942856
- [Background] Ritter MM, Sonnichsen AC, Mohrle W, Richter WO, Schwandt P. Beta-endorphin plasma levels and their dependence on gender during an enteral glucose load in lean subjects as well as in obese patients before and after weight reduction. Int J Obes. 1991 Jun;15(6):421-7. PMID 1885266
- [Background] Merchant RM, Yang L, Becker LB, Berg RA, Nadkarni V, Nichol G, Carr BG, Mitra N, Bradley SM, Abella BS, Groeneveld PW; American Heart Association Get With The Guidelines-Resuscitation Investigators. Incidence of treated cardiac arrest in hospitalized patients in the United States. Crit Care Med. 2011 Nov;39(11):2401-6. doi: 10.1097/CCM.0b013e3182257459. PMID 21705896
- [Background] Mulder M, Gibbs HG, Smith SW, Dhaliwal R, Scott NL, Sprenkle MD, Geocadin RG. Awakening and withdrawal of life-sustaining treatment in cardiac arrest survivors treated with therapeutic hypothermia*. Crit Care Med. 2014 Dec;42(12):2493-9. doi: 10.1097/CCM.0000000000000540. PMID 25121961
- [Background] Nolan JP, Berg RA, Callaway CW, Morrison LJ, Nadkarni V, Perkins GD, Sandroni C, Skrifvars MB, Soar J, Sunde K, Cariou A. The present and future of cardiac arrest care: international experts reach out to caregivers and healthcare authorities. Intensive Care Med. 2018 Jun;44(6):823-832. doi: 10.1007/s00134-018-5230-9. Epub 2018 Jun 2. PMID 29860705
- [Background] Perman SM, Stanton E, Soar J, Berg RA, Donnino MW, Mikkelsen ME, Edelson DP, Churpek MM, Yang L, Merchant RM; American Heart Association's Get With the Guidelines(R)-Resuscitation (formerly the National Registry of Cardiopulmonary Resuscitation) Investigators. Location of In-Hospital Cardiac Arrest in the United States-Variability in Event Rate and Outcomes. J Am Heart Assoc. 2016 Sep 29;5(10):e003638. doi: 10.1161/JAHA.116.003638. PMID 27688235